CLINICAL TRIAL: NCT05183451
Title: Effect of Low-level Laser Therapy on the Rate of En-masse Retraction in Adult Females With Bimaxillary Dentoalveolar Protrusion: a Single-center Randomized Clinical Trial
Brief Title: Effect Of Low Level Laser Therapy on the Rate of En- Masse Retraction: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Mohamed El- Sayed Dehis, Lecturer of Orthodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDCU-REC (2)/12-2018
Record Dates: First submitted 2021-12-05; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Bimaxillary Protrusion
Keywords: En-masse retraction; Rate of tooth movement; Low Level Laser Therapy (LLLT); 3D
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention neither the operator nor the patients could be blinded. The assessors will be blinded from the data to be investigated he will just measure the data needed without knowing the purpose of the study, and without knowing which records belong to which group. Two assessors will carry out the the analysis of the study, blindly and independently.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LG (Group A) (Experimental): En- masse retraction using NiTi closed coil springs rendering 200 g/side were employed following first premolars extraction and insertion of buccal TADs to provide maximum anchorage. Retraction was done along with the application of LLLT till the end of retraction.
  Interventions: Procedure: En- masse retraction and LLLT
- NLG (Group B) (Active Comparator): En- masse retraction using NiTi closed coil springs rendering 200 g/side were employed following first premolars extraction and insertion of buccal TADs to provide maximum anchorage. No LLLT was applied to this group
  Interventions: Procedure: En- masse retraction without LLLT

INTERVENTIONS:
Procedure: En- masse retraction and LLLT — Retraction will start on a 0.019"x0.025" Stainless steel wire using NiTi closed coils (force applied will be 200 g per side) extending between the crimpable hooks and the TADs. LLLT will be applied on days 0,3,7,14 from extraction then repeated biweekly till the end of retraction.
  Other Names: Laser group; Group A
  Arms: LG (Group A)
Procedure: En- masse retraction without LLLT — Retraction will start on a 0.019"x0.025" Stainless steel wire using NiTi closed coils (force applied will be 200 g per side) extending between the crimpable hooks and the TADs.
  Other Names: No laser group; Group B
  Arms: NLG (Group B)

SUMMARY:
There is scarcity in the literature regrading the effect of Low Level Laser Therapy (LLLT) on the rate of en-masse retraction. This study aims to investigate whether LLLT would affect the rate of en-masse retraction in females having bimaxillary dento-alveolar protrusion.

DETAILED DESCRIPTION:
Individuals having bimaxillary dentoalveolar protrusion are characterized by proclined upper and lower incisors and increased procumbency of the lips thus suffering from poor facial esthetics. The conventional management of these patients is the extraction of the first premolars and retraction of the anterior teeth.

One of the treatment techniques is in the form of canine retraction followed by four incisors retraction. This conventional method takes tedious work and tremendous time, thus affecting the patients' satisfaction adversely. The other technique is retraction of the whole set of anterior teeth as one unit (Canine and incisors), which is referred to as "En-Masse retraction".

Enhancing the rate of orthodontic tooth movement has always been a supreme goal of orthodontic research hoping to raise the level of care delivered to patients, hence, increase patients' satisfaction.

One of the proposed modalities of increasing the rate of tooth movement is Low Level Laser Therapy (LLLT). Thus, the aim of the current consideration was to evaluate the impact of LLLT on the rate of en-masse retraction in adult females having bimaxillary dentoalveolar protrusion.

ELIGIBILITY:
Inclusion Criteria:

* Adult females
* Patients having bimaxillary dento- alveolar protrusion and Class I Molar relation
* Cases requiring maximum anchorage during retraction.
* Good general and oral health

Exclusion Criteria:

* Patients suffering from any systemic diseases interfering with tooth movement.
* Patients with extracted or missing permanent teeth. (except for third molars).
* Patients with badly decayed teeth (Other than 1st premolars).
* Patients with any parafunctional habits (i.e. Bruxism, tongue thrusting, mouth breathing, etc…).
* Patients with previous orthodontic treatment
* Pregnant females

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-12-02 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Rate of en-masse retraction | From date of first premolars' extraction until the date of anterior teeth retraction, assessed up to an average of 1 year
  The antero-posterior movement of anterior teeth will be assessed by measuring the digitilized study models taken of the patients monthly (measured in mm)

SECONDARY OUTCOMES:
Anterior teeth's root resorption | From date of first premolars' extraction until the date of anterior teeth retraction, assessed up to an average of 1 year
  Assessed via comparing the pre & post- retraction CBCTs using Lavender & Malmgren Grading system
Anterior teeth Tip and Torque | From date of first premolars' extraction until the date of anterior teeth retraction, assessed up to an average of 1 year
  By comparing angular changes in the teeth's tip and torque in relation to reference planes
Anchorage (Loss/ Gain) | From date of first premolars' extraction until the date of anterior teeth retraction, assessed up to an average of 1 year
  By comparing linear and angular changes in the first molars in relation to reference planes
First molars' rotation | From date of first premolars' extraction until the date of anterior teeth retraction, assessed up to an average of 1 year
  Study models that are taken pre and post retraction (then digitilized) will be used to assess the rotation of the maxillary first molars in relation to a reference line
Pain Associated | From date of first premolars' extraction until the date of anterior teeth retraction, assessed up to an average of 1 year
  Each patient will fill a questionnaire regarding his treatment experience in a VAS scoring from 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Heba Mohamed E Dehis, Lecturer, Principal Investigator — Cairo University; Foad A El-Sharaby, A. Professor, Study Director — Cairo University; Faten H Eid, Professor, Study Director — Cairo University; Mushira Dahaba, Professor, Study Director — Cairo University; Yehya A Mostafa, Professor, Study Director — Future University in Egypt (FUE)
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Research data will be available for researchers who provide a methodologically sound proposal.
  Proposals should be directed to the corresponding author. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available immediately following publication and ending 6 months following article publication
Access Criteria: Data will be available after contact with the corresponding author
URL: https://fsharaby@hotmail.com

REFERENCES:
- [Derived] Dehis HM, El Sharaby FA, Eid FH, Mostafa YA. Effect of low-level laser therapy on en masse retraction in females with bimaxillary dentoalveolar protrusion : A single-center randomized clinical trial. J Orofac Orthop. 2025 Sep;86(5):284-297. doi: 10.1007/s00056-024-00525-2. Epub 2024 Jun 6. PMID 38842738